CLINICAL TRIAL: NCT06228300
Title: Registro Italiano Dei Pazienti Affetti da Dolore Cronico
Acronym: REALIZER
Status: Not yet recruiting | Type: Observational
Sponsor: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Responsible Party: Principal Investigator, Silvia Natoli, Principal Investigator, Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva
Other Study IDs: REALIZER
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Invasive pain management; Medical Pain Managemnet
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this Multicenter, non-profit, noninterventional, prospective observational cohort study is to create a register of patients suffering from Chronic Pain of any origin in subject with diagnosis of Chronic Pain according to the IASP19 criteria (Subjects > 4 years old - NRS > 4)

The main question[s] it aims to answer are:

Identify the profiles of patients belonging to pain therapy centers Evaluate the proportion of patients who reach the outcome of 30 or 50% improvement Evaluate the healthcare resources used in terms of number of accesses and time needed to achieve the best outcome (30 or 50% improvement) Identify patient profiles in terms of clinically significant outcomes in relation to baseline characteristics and specific treatments performed and their intermediate surrogate outcomes in relation to specific patterns Describe the relevant clinical variables in the study population. In particular, the absolute and relative frequencies of those clinical variables relevant to the effectiveness of the treatment will be described, categorized by type of treatment, and the timing of the start of treatment with respect to the onset of pain. The data collected may be used for predictive analyses Participants with a diagnosis of chronic pain (pain lasting > 12 weeks) will be enrolled, regardless of the etiology, modality and age of onset.

DETAILED DESCRIPTION:
The study aims to collect demographic and clinical data from patients belonging to pain therapy centers recognized at the regional level and belonging to the pain therapy networks established incompliance with law 38/2010 and according to the Agreement between the Government and the Regions of 25 July 2012.

Patients will be registered regardless of the access modality (outpatient or hospitalization) and will be characterized by pathology and treatments performed. The participation of centers for the treatment of pediatric pain is expected. Data relating to patients under the age of 18 will be analyzed separately.

The database aims to follow the patients enrolled according to a code that makes them anonymous.

Participating Centers The dissemination phase constitutes an integral part of the study and is not possible to predict the definitive number of centers involved. Key professionals have been contacted who will be responsible for the dissemination and implementation of this study based on each center's records. The ethics committee of the coordinating center will be regularly updated by the Principal Investigator as new centers join the study.

STUDY POPULATION The Registry data will be collected by the structures involved in the management of patients suffering from chronic pain, regardless of the cause. It is necessary to keep the inclusion criteria as broad as possible to obtain a real picture of clinical practice at a national level.

Inclusion criteria

* Subjects > 4 years old
* NRS > 4
* Diagnosis of Chronic Pain according to the IASP19 criteria
* Adherence through written informed consent to participate in the study Exclusion criteria
* Patients suffering from psychiatric pathology or severe cognitive impairment for which the enrolling doctor does not believe it is useful for the purposes of the study
* Patients unable to sign the informed consent Description of the pathologies being studied Adult and pediatric patients will be enrolled, diagnosed with Chronic Pain (pain lasting > 12 weeks), regardless of the etiology, modality, and age of onset.

PROCEDURES EXPECTED AND INFORMATION COLLECTED Enrollment procedure Adult and pediatric patients (> age 4) of both sexes who belong to pain therapy centers with a diagnosis of Chronic Pain (pain that lasts > 12 weeks), regardless of the etiology, modality and age of onset, will be considered eligible for enrollment.

Patients (or parents if pediatric) will be asked to join the study after having been informed in detail (also with the aid of a written information form) of the objectives of the project, as well as the methods with which these objectives will be pursued. Participants will be informed about the lack of informative feedback regarding the results of future clinical evaluations: the results of any research originating from the register, in fact, will not be delivered to the participants themselves. The subject who freely accepts will authorize the inclusion of their data in the project by signing the informed consent form of which they will receive a copy. It will also be clearly explained in the information sheet attached to the informed consent that each participant will have the possibility of withdrawing their participation from the study at any time, without providing any reason and without this jeopardizing the doctor-patient relationship with the specialists involved in the project.

Patients will be informed by the manager of the patient's pain center or the principal investigator for the center (assuming this is not the same individual).

The doctor will complete the electronic CRF after evaluating the patient and classifying him according to the criteria of the IASP (International Association for the Study of Pain) in terms of primary or secondary chronic pain. In the case of a patient enrolled during a check-up or during hospitalization, all data relating to the time in which the patient is in care at the center, the invasive procedures previously undertaken, the drugs prescribed, will be collected. Retrospective data (only for patients already being treated at the center) will be collected according to a predefined group (e.g.: the patient has been in the care of the center for: > 5 years; from 1 to 5 years; from 1 year to 6 months; from 3 to 6 months; < 3 months).

Follow-up procedure Once enrolled, the patient will be followed prospectively until the end of enrollment. At each visit it will be possible to retrieve the patient's chart and fill in the data relating to the intensity of pain and the treatments undertaken. It will also be possible to modify or add an etiological diagnosis in forms of secondary chronic pain. There is no limit to the number of follow-ups for each patient as long as the database is active (3 months from the date of enrollment of the last patient, considering a 12-month active enrollment expected for this study).

Data gathered The activities of the registry do not replace routine diagnostic tests or visits to your doctor. The data collected by the registry will include relevant demographic data of the patient, comorbidities, the duration of the pain (> 5 years; from 1 to 5 years; from 1 year to 6 months; from 3 to 6 months), the type of pain, the location of the pain, the intensity of the pain (Brief Pain Inventory- Severity (BPI-S) and pain interference in daily activities (Brief Pain Inventory- Interference (BPI-I), treatments received (categorized according to pharmacological therapy, infiltrative therapy, ablative or neuromodulatory therapy, implants), the tests conducted, the number of other medical specialists contacted for the pathology being studied, the professional who sent it to the center.

In particular, patients will be characterized by:

Location of pain according to the following scheme (multiple options are possible) Lower back pain Thoracic Upper arts Lower limbs Head/Neck Pelvis Pain Intensity Brief Pain Inventory-Severity (BPI-S) Interference with daily activities Brief Pain Inventory-Interference (BPI-I) Clinical information related to the pathology Therapy Pharmacological Infiltrative Mini-invasive Implantable Data collection methods and anonymization The data collected will be used for scientific and epidemiological purposes. Each data will be created by a participating center and recorded on the SIAARTI Servers via a web application using the RedCap® data management software.

The study data will be collected and managed using the REDCap2electronic data acquisition tools made available by SIAARTI. REDCap (Research Electronic Data Capture) is a secure, web-based software platform designed to support data capture for research studies. It provides:

1. an intuitive interface for acquiring validated data;
2. Controlled channels with customized access privileges for monitoring data manipulation and export procedures;
3. automated export procedures for continuous data download to common packages of statistical software;
4. procedures for data integration and interoperability with external sources. Data will be recorded in the e-CRF only after being anonymized using coding procedures described in a separate document, in accordance with applicable data protection laws, including the EU GDPR. The encryption key of the anonymous data which contains the patient's name, surname and date of birth will be archived only in the files of the local site in a register that allows registration and research of the subject.

For each center participating in the project, an account will be created on the REDCap platform. The data will be recorded using an encrypted data connection (HTTPS) of anonymized input via a web browser or mobile app.

To enable data analysis, each patient will be assigned a unique Subject ID (Patient Identification Number).

REDCap is a secure web application for creating and managing online databases. Unauthorized access to data is impossible since access is permitted according to a hierarchical and role-based criterion. Access to REDCap will be allowed only to data collection personnel of the participating centers, according to the methods established by this protocol. These people will keep the information private.

Data management and storage RedCap management software will be used for data management. The identification of individual patients by name will not be necessary or required at any time. During the collection and processing of data, therefore, all necessary measures will be adopted to effectively establish anonymization. SIAARTI will also take care of data storage. Each participating center can only access the patient data it has generated and registered on the REDCap platform. Each participating center is required to provide periodic ad hoc reports on the data collected.

Data ownership Individual data provided by a participating center are primarily the property of the center that generated the data. All investigators have the right to access their data at any time. SIAARTI will be co-owner of the data, in agreement with each participating center.

Subsequent use of the data SIAARTI and the executive committee, on behalf of the investigators, have the right to use all data collected in the database for scientific purposes. The executive committee and the SIAARTI study groups have the right to access the data in the registry, for research purposes after the conclusion of the research project, and with the approval of the SIAARTI Scientific Committee. In any case, the researchers who contributed to the project will be regularly informed about the ongoing study activities and will be given the opportunity to be included among the authors of any publications.

Storage A copy of the electronic database will be kept at the SIAARTI headquarters and kept for 5 years for subsequent use by SIAARTI and the executive committee.

ENDPOINT Primary Endpoint The number of patients referring to the centers, the type of pain, the proportion of patients who reach the clinically significant outcome, the type of therapies prescribed (pharmacological, neuromodulatory or implanted) necessary to achieve the outcome and the number of accesses and the Time in which a clinically significant improvement will be achieved (Change in BPI-s or BPI-I; a reduction of > 30% is considered clinically significant and a reduction of > 50% is considered optimal, the data will be evaluated for each Item).

Secondary Endpoint

1. The effectiveness of the treatments will be described in terms of

   1. Change in pain intensity according to the Brief Pain Inventory-Severity questionnaire (BPI-S) A reduction of > 30% is considered clinically significant and optimal a reduction > of 50% the data will be evaluated for each Item)
   2. b. Change in pain interference on daily activities according to the Brief Pain Inventory-Interference questionnaire (BPI-I). A reduction of > 30% is considered clinically significant and a reduction of > 50% is considered optimal; the data will be evaluated for each item)
2. Proportion of patients achieving clinically significant outcomes in relation to baseline characteristics and specific treatments performed and their intermediate surrogate outcomes in relation to specific patterns.
3. Resources used: Number of visits to the center for each patient in a year; Number of ordinary or day hospitalizations for each patient in a year.
4. The clinical variables relevant to the outcome will be described (e.g. type of pain, comorbidities, the time between treatment and clinically significant improvement, type of therapy undertaken - pharmacological, invasive, implant-based) INFORMED CONSENT Patients enrolled in the study will be given a complete and exhaustive explanation about the nature, purposes, possible risks, and benefits of the study. The patient will be informed that he/she will be free to stop the study at any time. The patient will be given the opportunity to ask questions and will be given as much time as desired to evaluate the information provided. For the pediatric population, consent will be requested from parents in the same way.

The investigating doctor will keep the original of the signed written informed consent.

In the written informed consent form it will be specified that the study data will be stored in computerized form and that the confidentiality of the data itself will be maintained in accordance with the provisions of current legislation.

STATISTICAL ANALYSIS All enrolled patients registered in the registry will be included in the analyses. A descriptive analysis will be performed on the collected data. In general, qualitative variables will be described using frequency distributions; the quantitative variables will be described by mean and standard deviation if normally distributed, and by median and interquartile range if asymmetrically distributed. As appropriate, statistical tests will be used for exploratory purposes. Treatment effects (Change in BPI-S and BPI-I scores) will be calculated as the ratio of the difference between baseline and follow-up scores to the baseline score. If the data allow it, inferential analysis will be applied on quantitative data (such as: comparison of Student's t means, Fisher's F, etc.), or on qualitative data (such as: chi square, odds ratio, Mann Whitney U, etc.). The prevalence of the different pathologies and the related confidence intervals will be estimated. Detailed statistical analysis plans will be set up in future research protocols that will use this database as a source of data.

Sample Size Since this is an observational registry, no prior sample size calculation is required.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 4 years old
* NRS > 4 - Diagnosis of Chronic Pain according to the IASP19 criteria
* Accession through written informed consent to participate in the study

Exclusion Criteria:

* Patients suffering from psychiatric pathology or severe cognitive impairment for which the enrolling doctor does not believe it is useful for the purposes of the study;
* Patients unable to sign the informed consent.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients suffering from chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of the profile of patients admitted to pain clinics in Italy: number of patients admitted | one year
  Progressive count
Characterization of the profile of patients admitted to pain clinics in Italy: type of pain. | one year
  A semplified ICD-11 Classification will be used
Characterization of the profile of patients admitted to pain clinics in Italy: proportion of patients who reach a clinically significant outcome. ; time in which a clinically significant improvement will be achieved | one year
  The Brief Pain Inventory questionnaire will be used to assess efficacy of treatmens. 30% of reduction will be considered clinically relevant
Characterization of the profile of patients admitted to pain clinics in Italy: type of prescribed therapies (pharmacological, neuromodulatory or implant) necessary to achieve a clinically significant improvement | one year
  Description of treatments offered to each patient
Characterization of the profile of patients admitted to pain clinics in Italy: time in which a clinically significant improvement will be achieved | one year
  Number of days needed to reach a clinically relevant outcome

SECONDARY OUTCOMES:
Resources employed for each patient | one year
  Number of admissions and kynd of admissions (inpatient,outpatient)
Proportion of patients who reach an optimal improvemnet | one year
  Proportion of patients with more than 50% reduction of Brief Pain inventory score

DOCUMENTS (1):
  • Study Protocol (2022-10-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT06228300/Prot_000.pdf